CLINICAL TRIAL: NCT00853619
Title: Clinical Decision Support Consortium for AHRQ CDS Research
Brief Title: Clinical Decision Support Consortium
Acronym: CDSC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Blackford Middleton, MD, MPH, Study Principal Investigator, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HHSA290200810010
Record Dates: First submitted 2009-02-26; First posted 2009-03-02 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes; Coronary Artery Disease; Hypertension
Keywords: clinical decision support; knowledge management; knowledge representation; clinical guidelines; coronary artery disease; myocardial ischemia; diabetes mellitus; hypertension
MeSH Terms: conditions — Diabetes Mellitus; Coronary Artery Disease; Hypertension; Myocardial Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Services Demo at PHS and RI (Experimental): Service based CDS intervention at PHS.
  Interventions: Other: Service based decision support intervention
- Normal CDS interventions at PHS and RI (Active Comparator): Normal CDS intervention at both PHS and RI hospitals
  Interventions: Other: Service based decision support intervention

INTERVENTIONS:
Other: Service based decision support intervention — Delivering CDS via services
  Other Names: Clinical Decision Support,; CDS Consortium,; Enterprise Clinical Rules Services

SUMMARY:
The goal of the Clinical Decision Support (CDS) Consortium research study is to assess, define, demonstrate, and evaluate best practices for knowledge management (KM) and CDS in healthcare information technology across multiple ambulatory care settings and electronic health records (EHR) technology platforms.

There are seven specific research objectives focusing on two practical areas of implementation for clinical decision support services: a) healthcare maintenance and preventive care screening, and b) two chronic disease conditions: Coronary Artery Disease (CAD), and Adult-onset Diabetes Mellitus (AODM). The research objectives are: 1) Knowledge management lifecycle, 2) Knowledge specification, 3) Knowledge portal and repository, 4) CDS knowledge content and public web services, 5) CDS Dashboard, 6)Evaluation, and 7) Dissemination.

DETAILED DESCRIPTION:
Investigators and developers of electronic health records from both academe and industry have come together to form the Clinical Decision Support (CDS) Consortium. Members of the CDS Consortium are intimately involved in creating and providing CDS tools and services in electronic health records used in both academic settings as well as community-based physician office practices. These investigators share a common interest and goal of enhancing the wide-spread adoption of CDS tools and services to improve the delivery of healthcare both domestically and world-wide.

Our approach to the project is iterative and cyclical: we will begin with a survey of the knowledge management lifecycle and supporting infrastructure (such as knowledge management systems, terminology services and data standards) at the participating clinical sites. We will then work together to define best practices for translating knowledge into a multi-layered array of human readable knowledge artifacts and public web services. At each point in this process, we will conduct careful evaluation, documenting lessons learned from each site. The ultimate work products will fall into three main categories:

First, tangible, actionable knowledge artifacts such as the shareable, human-readable and computable forms of clinical practice guidelines (CPGs) under study, public web-services for CDS demonstrations, and a CDS Knowledge Portal and Repository to facilitate widespread adoption of these artifacts.

Second, detailed guidance and recommendations, based on what we learn from our combined efforts, for external parties such as the Certification Commission for Health Information Technology (CCHIT), the Health Information Technology Standards Panel (HITSP), and the clinical practice guideline developer community.

Third, a set of knowledge and best practices, such as methods for the knowledge management lifecycle, development of both human readable knowledge artifacts and machine-interpretable knowledge, and management of decision-support related organizational change. We will share this knowledge through a variety of channels, such as presentations and academic papers.

ELIGIBILITY:
Inclusion Criteria:

* PHS clinics using the LMR (Partners electronic health record system). These clinics include Massachusetts General Hospital Back Bay, Brigham Primary Physicians at Faulkner Hospital, Brigham PCA in Brookline, and Brigham and Women's Hospital at Foxboro.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2008-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Compliance with guideline | 6 months

SECONDARY OUTCOMES:
Patient outcomes | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Blackford Middleton, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Partners HealthCare - Information Systems, Wellesley Gateway, Wellesley, Massachusetts, United States

REFERENCES:
- [Background] Middleton B. The clinical decision support consortium. Stud Health Technol Inform. 2009;150:26-30. PMID 19745260
- See also: Clinical Decision Support Consortium Website — http://www.partners.org/cird/cdsc